CLINICAL TRIAL: NCT06143007
Title: A Phase I, Open-label, Multicenter Study to Assess Safety, Tolerability, Pharmacokinetic, Efficacy and Preliminary Food Effect of BB3008 Tablet Administered Orally to Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of BB3008 in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Broadenbio Ltd., Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB3008-ST-I-02
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
Keywords: BB3008; HPK1; First-in-Human; Dose Escalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BB3008 monotherapy (Experimental): The study is composed of fasted dose cohorts and fed dose cohort. BB3008 will be administered orally daily alone as monotherapy in all cohorts. In the fasted dose cohorts, the subjects will receive once daily of BB3008 monotherapy fasted across approximately 6 ascending dose levels. The starting dose is 80 mg/day. In the fed dose cohort, the subjects will receive once daily of BB3008 monotherapy in a fed condition. The dose selected for fed dose cohort must be deemed safe as assessed by safety monitoring committee (SMC).
  Interventions: Drug: BB3008 tablet

INTERVENTIONS:
Drug: BB3008 tablet — BB3008 tablets will be administered orally once daily (QD).
  Other Names: BB3008

SUMMARY:
This is a Phase 1 dose escalation study to evaluate the safety, tolerability, pharmacokinetics, efficacy and preliminary food effect of BB3008 as monotherapy in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This first-in-human (FIH) study of BB3008 will evaluate safety, tolerability, pharmacokinetics (PK) efficacy and preliminary food effect of BB3008 in subjects with advanced solid tumors. The primary objective is to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of BB3008 as monotherapy, and to evaluate the safety and tolerability of BB3008. The secondary objectives include the assessments of PK profile, preliminary efficacy, preliminary food effect (FE) and preliminary metabolites identification of BB3008. The exploratory objectives are to explore biomarkers and C-QTcF analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed of the study and voluntarily signed the informed consent form (ICF), and willing to follow and have the ability to complete all trial procedures.
2. Subjects with histologically or cytologically confirmed advanced solid tumors who are lacking standard therapy, progressing after adequate standard therapy, or intolerant of standard therapy.
3. ECOG score ≤1.
4. At least one evaluable or measurable lesion as defined by RECIST v1.1.
5. Expected survival ≥ 3 months.
6. adequate organ function.
7. Female subjects of childbearing potential must have a negative pregnancy test prior to the first dose and are required to use effective contraception from signing the ICF until 6 months after the last dose of study treatment.

Exclusion Criteria:

1. History of dual-source cancer within 5 years.
2. Presence of known active central nervous system (CNS) and/or leptomeningeal metastases.
3. History of clinically serious cardiovascular and cerebrovascular disease within 6 months.
4. Active infection (including, but not limited to HBV or HCV).
5. Received radical radiotherapy within 12 weeks.
6. Received live virus vaccination within 4 weeks.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | Single dose to the end of Cycle 1 (each cycle is 21 days)
  To assess the safety and tolerability of BB3008 tablet as monotherapy in subjects with advanced solid tumors and to determine the maximum tolerated dose (MTD) of BB3008 tablet, and to provide a basis for determination of the recommended dose (RP2D) for Phase II clinical trials.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28 to Day -1) through up to 12 months or until disease progression
  AEs and SAEs will be characterized by type, seriousness, relationship to study treatment, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) and timing.

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: Peak Plasma Concentration (Cmax) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Time to Peak Concentration (Tmax) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Area under the plasma concentration-time curve (AUC) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Pharmacokinetic Assessments: Elimination half-life (t½) | Day 1, Day 8, Day 15 and at the end of Cycle 1 (each cycle is 21 days)
  Blood samples will be collected for PK analyses
Objective response rate (ORR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Duration of response (DOR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Disease control rate (DCR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.
Progression-free survival (PFS) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality